CLINICAL TRIAL: NCT04999553
Title: Left Intermittent Theta Burst Stimulation vs. Right Low Frequency Repetitive Transcranial Magnetic Stimulation Effectiveness in Depression and Suicidal Ideation: A Randomized Non-Inferiority Trial
Brief Title: Left vs. Right Non-Inferiority Trial
Acronym: LeRNIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-00583
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Depression; Major Depressive Disorder; Major Depressive Episode
Keywords: rTMS; TMS; Transcranial Magnetic Stimulation; iTBS; Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a two-arm multicenter parallel, clinician-blinded randomized non-inferiority trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study doctors and raters obtaining outcome measures will be blind to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Theta Burst Stimulation (iTBS) (Active Comparator): iTBS to the L-DLPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Intermittent Theta Burst Stimulation (iTBS)
- Low Frequency Right (LFR) (Active Comparator): 1Hz stimulation to the R-DLPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Low Frequency Right (LFR)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS will employ the MagPro X100/R30 stimulator equipped with the cool-B70 as we used a cool-B70 in our past non-inferiority trial. The dose will be a 120% rMT in accordance to our latest trial using iTBS. The target area to stimulate will be the right dorsolateral prefrontal cortex (DLPFC) for LFR and the left DLPFC for iTBS as established in prior clinical trials. The localization of both targets will follow the well-established procedures for either R-DLPFC or L-DLPFC using a heuristic method.
Device: Intermittent Theta Burst Stimulation (iTBS) — Intermittent Theta Burst Stimulation (iTBS)
  Arms: Intermittent Theta Burst Stimulation (iTBS)
Device: Low Frequency Right (LFR) — Low Frequency Right (LFR)
  Arms: Low Frequency Right (LFR)

SUMMARY:
The aim of this study is to test the hypothesis that low-frequency rTMS (LFR) works as well as the established intermittent thetaburst rTMS (iTBS) treatment for treatment resistant depression (TRD).

DETAILED DESCRIPTION:
In this multi-centre, triple-blinded, non-inferiority trial 420 patients with TRD will be recruited at two academic centres (UBC, CAMH). Patients will be randomised to receive either iTBS or LFR for 30 sessions. The primary outcome will be the improvement on a depression scale. Secondary outcome will be improvement of suicidal ideation. A secondary aim is to test the predictive capacity of a novel, easy to implement heart rate based biomarkers (i.e. heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

1. are female or male;
2. are outpatients;
3. are voluntary and competent to consent to treatment;
4. have a DSM 5 diagnosis of MDD,55 single or recurrent confirmed by Mini-International Neuropsychiatric Interview (MINI) version 7.0;
5. are 18yo to 65yo;
6. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode OR have been unable to tolerate at least two separate trials of antidepressants at less than the minimum adequate dose and/or duration (ATHF 1 or 2);
7. have a score ≥ 18 on the Hamilton Depression Rating Scale (HDRS-17 item);
8. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening;
9. are able to adhere to the treatment schedule;
10. pass the TMS and MRI adult safety screening questionnaires.

Exclusion Criteria:

1. have a history of substance use within the last 3 months;
2. have a concomitant major unstable medical illness;
3. have active suicidal intent;
4. are pregnant;
5. have a lifetime (MINI) diagnosis of any psychotic or bipolar disorder;
6. have a MINI anxiety disorder or personality disorder assessed by a study investigator to be primary and causing greater impairment than MDD;
7. have failed a course of ECT in the current episode;
8. have any significant neurological disorder, any history of seizure (except those therapeutically induced by ECT), significant head trauma with loss of consciousness for > 5 min;
9. have any intracranial implant (e.g., aneurysm clips) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
10. are participating in psychotherapy, must have been in stable treatment for at least 3 months prior to study entry, with no anticipated change in the frequency of therapeutic sessions, or focus of therapeutic sessions over the duration of the study;
11. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
12. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 30 days
  17 item Hamilton Depression Rating Scale (HDRS-17) Change

SECONDARY OUTCOMES:
Suicidal ideation | 30 days
  Columbia Suicide Severity Rating Scale Screen Version (C-SSRS) Change
Anxiety severity | 30 days
  Hamilton Anxiety Rating Scale (HAM-A) Change
Depression severity | 30 days
  Self-rated 16-item Quick Inventory of Depressive Symptoms (QIDS-16) Change

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Non-Invasive Neurostimulation Therapies Centre, University of British Columbia, Vancouver, British Columbia
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No